CLINICAL TRIAL: NCT00004149
Title: A Phase II Trial of Arsenic Trioxide in Advanced Hormone-Refractory Prostate Cancer
Brief Title: Arsenic Trioxide in Treating Patients With Stage IV Prostate Cancer That Has Not Responded to Previous Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Model: Parallel | Purpose: Treatment
Other Study IDs: CDR0000067382; AECM-1199908270; NCI-T99-0077; AECM-CCRC-9929
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Prostate Cancer
Keywords: stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Arsenic Trioxide

INTERVENTIONS:
Drug: arsenic trioxide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of arsenic trioxide in treating patients who have stage IV prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of arsenic trioxide in patients with metastatic stage IVA or IVB hormone-refractory prostate cancer.
* Determine the toxicity of this drug in this patient population.
* Assess, in a preliminary manner, the effect of this drug on pain control in these patients.
* Assess the potential value of serial quantitative prostate-specific antigen (PSA) and prostate-specific membrane antigen (PSMA) mRNA determinations in RNA from peripheral blood mononuclear cells as surrogate markers of disease response in patients treated with this drug.
* Assess the pharmacokinetics and pharmacodynamics of this drug in these patients.
* Assess the feasibility of using pretreatment bone marrow evaluation of PSA and PMSA mRNA levels and pi class glutathione S-transferase expression (i.e., eliminate glutathione levels) as potential correlates of disease response in patients treated with this drug.

OUTLINE: Patients receive arsenic trioxide IV over 2 hours on days 1-5 and 8-12 for one course. Treatment continues as biweekly infusions for at least 14 additional weeks in the absence of disease progression, unacceptable toxicity, or excessive increase in serum prostate-specific antigen.

Pain is assessed at baseline and then before each biweekly treatment.

PROJECTED ACCRUAL: A total of 17-37 patients will be accrued for this study within 12-24 months.

ELIGIBILITY:
Eligibility Criteria:

* Diagnosis of stage IVA or IVB hormone-refractory prostate cancer
* Obstructive uropathy and/or hydronephrosis allowed if adequate renal function and urinary drainage
* WBC at least 2,500/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9.0 g/dL
* Bilirubin less than 2 mg/dL

Exclusion Criteria:

* No significant active infectious disease
* No grade 2 or greater peripheral neuropathy
* No other debilitating acute or chronic co-morbid medical, neurological, or psychiatric condition that would preclude study compliance
* No concurrent amphotericin B or other agent that prevents restoration of potassium or magnesium to normal levels and/or correction of QT interval to under 500 milliseconds

Max Age: 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 1999-09 (Actual); Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert E. Gallagher, MD, Study Chair — Albert Einstein College of Medicine
Locations (3):
- United States (3):
  - Mount Sinai Medical Center, NY, New York, New York
  - Jacobi Medical Center, The Bronx, New York
  - Albert Einstein Clinical Cancer Center, The Bronx, New York

REFERENCES:
- [Result] Gallagher RE, Ferrari A, Kaubisch A, et al.: Arsenic trioxide (ATO) in metastatic hormone-refractory prostate cancer (HRPC): results of phase II trial T99-0077. [Abstract] J Clin Oncol 22 (Suppl 14): A-4638, 2004.